CLINICAL TRIAL: NCT00045526
Title: Phase II Study Of OSI-774 In Advanced Esophageal Cancer
Brief Title: Erlotinib Hydrochloride in Treating Patients With Advanced Esophageal Cancer or Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01418; 02-035; NSC-718781; NCI-5445; CDR0000256601; MSKCC-02035; N01CM62206 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Recurrent Esophageal Cancer; Squamous Cell Carcinoma of the Esophagus; Stage III Esophageal Cancer; Stage IV Esophageal Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying erlotinib hydrochloride to see how well it works in treating patients with advanced esophageal cancer or stomach cancer. Erlotinib hydrochloride may stop the growth of cancer by blocking the enzymes necessary for tumor cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with advanced carcinoma of the esophagus or gastroesophageal junction treated with erlotinib (erlotinib hydrochloride).

II. Determine the overall survival of patients treated with this drug. III. Determine the degree of dysphagia relief in patients treated with this drug.

IV. Determine the toxicity and tolerability of this drug in these patients. V. Correlate epidermal growth factor receptor (EGFR) expression with response to treatment in these patients.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once daily (QD). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma, squamous cell or small cell carcinoma, or carcinoma not otherwise specified of the esophagus or gastroesophageal junction

  * Metastatic or surgically unresectable disease
* Measurable disease outside of primary tumor

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral computed tomography (CT) scan
* No bone metastases, abnormal radionuclide bone scans, or pleural effusions as only site of measurable disease
* No known brain metastases or carcinomatous meningitis
* Must consent to having tumor tissue tested for epidermal growth factor receptor status
* Performance status-Karnofsky 70-100%
* Life expectancy of greater than 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) no greater than 2 times ULN
* Creatinine no greater than 1.5 mg/dL
* Calcium no greater than 12 mg/dL
* No symptomatic hypercalcemia
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No ventricular arrhythmia
* No other malignancy within the past 3 years except adequately treated carcinoma in situ of the cervix, superficial transitional cell carcinoma of the bladder, or basal cell or squamous cell skin cancer
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No other concurrent disease that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior cetuximab
* No more than 1 prior chemotherapy regimen for advanced or metastatic disease
* One prior chemotherapy in the adjuvant setting (in combination with prior surgery or radiotherapy) allowed provided it was administered prior to treatment for advanced or metastatic disease
* At least 3 weeks since prior chemotherapy
* No concurrent investigational or commercial chemotherapy
* At least 3 weeks since prior radiotherapy
* No prior erlotinib-related compounds or compounds of similar biologic or chemical components
* No prior EGFR-targeting compounds (e.g., gefitinib)
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2002-06; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Major response rate (complete and partial response) | Up to 5 years

SECONDARY OUTCOMES:
Toxicities, graded according to the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) | Up to 5 years
Degree of dysphagia relief | Up to 5 years
Time to progression | Up to 5 years
  Estimated using the Kaplan-Meier method and confidence intervals will be formed for median time to progression.
Overall survival | Up to 5 years
  Estimated using the Kaplan-Meier method and confidence intervals will be formed for median survival time.

CONTACTS AND LOCATIONS:
Overall Officials: David Ilson, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States